CLINICAL TRIAL: NCT04675281
Title: Pathological Findings in Critically-ill Patients Who Died From SARS-CoV-2 Related Acute Respiratory Distress Syndrome
Brief Title: Pathological Findings of Fatal COVID-19
Acronym: HISTOCOVID
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: MR_HISTOCOVID
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: SARS-CoV-2; Covid19; Pathology; Intensive Care Units; Respiratory Distress Syndrome
Keywords: SARS-CoV-2; Pneumonia; Intensive care units; Acute Respiratory Distress Syndrome; Histopathology
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lung biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically-ill adult patients who died in the Intensive Care Unit from a documented COVID-19
  Interventions: Other: 2 post-mortem transcutaneous lung biopsies (1 anterior ; 1 posterior) using anatomical landmarks

INTERVENTIONS:
Other: 2 post-mortem transcutaneous lung biopsies (1 anterior ; 1 posterior) using anatomical landmarks — All specimens are fixed with 4% neutral formaldehyde and embedded in paraffin wax in the department of pathology of each participating centre. Afterwards, all samples are sent for analysis to the department of pathology of Nantes university hospital. All biopsies are independently analysed by a group of pathologists who are experts in lung tissue and blinded to clinical information. All biopsies will be analysed using a predetermined semi-quantitative histological scoring grid. The pathologists are asked to assess the degree of: edema, cell necrosis, hyaline membrane formation, proliferation of alveolar type 2 cells, fibrosis, capillary congestion, alveolar edema, neutrophilic infiltration, and microscopic thrombosis. Finally, the following patterns are recorded: exudative diffuse alveolar damage (DAD), proliferative DAD, fibrosis, intra-alveolar haemorrhage, lymphocytic pneumonia, organizing pneumonia, acute fibrinous organizing pneumonia (AFOP), thrombotic microangiopathy.

SUMMARY:
The Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) is a new coronavirus discovered in December 2019 in Wuhan, China and currently responsible of a worldwide outbreak and the death of more than 55,000 patients in France. The more severe form of COVID-19 disease induces a pneumonia with profound hypoxemia which may require invasive mechanical ventilation. It is estimated that 5% of COVID-19 patients are admitted to the Intensive Care Unit (ICU) for management. Hospital mortality in patients who develop severe acute respiratory distress syndrome (ARDS) ranges between 40% and 60%. The investigators purpose to investigate the pathological findings of COVID-19 patients who died from ARDS in the ICU by doing post-mortem lung biopsies

DETAILED DESCRIPTION:
Forty-four French ICUs participate to this study with the aim to perform 200 lung biopsies in 100 patients over a 12-month period. This cohort will be the largest pathological database of COVID-19 patients who developed ARDS. In accordance with the French law, this study has been approved and registered by the French Agency of Biomedicine and the French Ministry of Education and Research (#PFS 20-016). Two transcutaneous lung biopsies per patient will be performed using a 14G needle and anatomical landmarks (1 anterior biopsy and 1 posterior biopsy). All biopsies will be referred to the Department of Pathology of Nantes university hospital and analysed by a group of pathologists specialized in lung tissue. The primary objective is to describe and characterize the lesions of the lung induced by the SARS-CoV-2 infection. The secondary objectives are to correlate the pathological findings with the patients' demographics, the treatments administered during the ICU stay, the ventilator settings, to document the percentage of co-infections and their types, compare the radiographic findings (Chest X-ray and CT-scan of the chest) with the pathological findings, to compare the pathological findings of early deaths (<1week after ICU admission) versus late deaths (>1 week). These pathological findings will undoubtedly help to better understand the pathophysiology of SARS-CoV-2 pneumonia and pave the way to the development of new therapeutic strategies

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (Age≥18 years-old)
* Hospitalized in Intensive Care Unit (ICU)
* Dead in the ICU from documented Covid-19 (clinical and radiological signs of pneumonia with a positive SARS-Cov-2 PCR from the upper or lower respiratory tract)
* Not registered in the national register of refusal of the French Biomedicine Agency
* According to French law, there was no requirement for signed consent, but the patient's next of kin were informed about the study before enrolment and were given a letter of information about the study.

Exclusion Criteria:

* Covid-19 not documented by a positive SARS-Cov-2 PCR
* Patient with a positive SARS-Cov-2 PCR but without any signs of pneumonia during the ICU stay (no clinical and no radiological signs of pneumonia)
* Patient registered in the "national register of refusal" of the French Biomedicine Agency
* Refusal expressed by the patient's next of kin to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients deceased in the ICU from a Covid-19 during the study period
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Analysis of the pathological findings of a large cohort of patients who died from COVID-19 in the ICU | Two post-mortem lung biopsies performed immediately after death.
  Detailed description and analysis of the primary lesions of the lungs in patients who died in the ICU from Covid-19.

SECONDARY OUTCOMES:
Comparison between early (<1 week after ICU admission) and late (≥1 week) deaths | Two post-mortem lung biopsies performed immediately after death.
  Comparison of pathological findings according to the time between ICU admission and death.
Analysis of the influence of ARDS severity and length on pathological findings | Two post-mortem lung biopsies performed immediately after death.
  Comparison of pathological findings according to the length of acute respiratory syndrome.
Analysis of the influence of ARDS severity and length on pathological findings | Two post-mortem lung biopsies performed immediately after death.
  Comparison of pathological findings according to the duration of acute respiratory syndrome.
Analysis of the influence of pharmacological treatments (steroids) on pathological findings | Two post-mortem lung biopsies performed immediately after death.
  Comparison of pathological findings between patients who received steroids and those who did not.
Analysis of the correlation between radiological findings and pathological findings | Two post-mortem lung biopsies performed immediately after death.
  Comparison between radiological description of the CT of the lungs and the radiological findings.
Association between the primary cause of death and pathological findings | Two post-mortem lung biopsies performed immediately after death.
  Analysis of the pathological findings according to the primary cause of death (hypoxia, shock, hypoxia and shock, cardiac arrest, other).
Analysis of the correlation between the ventilator settings and pathological findings | Two post-mortem lung biopsies performed immediately after death.
  Analysis of the correlation between the ventilator settings (tidal volume, PEEP, driving pressure, plateau pressure, static compliance, volume or pressure mode) and pathological findings.
Co-infections | Two post-mortem lung biopsies performed immediately after death.
  Description of the co-infection (bacterial or fungal infections) documented by pathological findings

CONTACTS AND LOCATIONS:
Locations (44):
- France (44):
  - CH Amiens, Amiens
  - Angers University Hospital, Angers
  - CH Angoulême, Angoulême
  - CH Annecy, Annecy
  - Hopital Privé d'Antony, Antony
  - CH Argenteuil, Argenteuil
  - CH Belfort, Belfort
  - CHU Bordeaux, Bordeaux
  - Hopital Sainte Camille, Bry-sur-Marne
  - CH Cahors, Cahors
  - CH Cergy Pontoise, Cergy-Pontoise
  - CH Cholet, Cholet
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CH Compiègne-Noyon, Compiègne
  - CHD Vendée, La Roche-sur-Yon
  - Hopital Lyon Sud, Lyon
  - Hôpital Lyon Sud, Lyon
  - Marseille Hopital Nord APHM, Marseillette
  - CH Melun, Melun
  - CH Montélimar, Montélimar
  - Nantes University Hospital, Nantes
  - CHU Nice, Nice
  - CHR Orléans, Orléans
  - CH Ambroise Paré APHP, Paris
  - GHEF Marne La Vallée, Paris
  - Hopital Antoine Béclère APHP, Paris
  - Hopital Cochin APHP, Paris
  - Hopital Georges Pompidou APHP, Paris
  - Hopital La Pitié Salpetrière APHP, Paris
  - Hopital Louis Mourier APHP, Paris
  - Hopital Necker APHP, Paris
  - Hopital Saint-Antoine APHP, Paris
  - Hopital Saint-Louis APHP, Paris
  - CH Poissy, Poissy
  - Hopital Privé Claude Galien, Quincy-sous-Sénart
  - CH Reims, Reims
  - CHU Rennes, Rennes
  - CH Saint-Brieuc, Saint-Brieuc
  - CHU Saint-Etienne, Saint-Etienne
  - Hopital Foch, Suresnes
  - CHRU Tours, Tours
  - CH Troyes, Troyes
  - CH Vannes, Vannes
  - CH Versailles, Versailles

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Morin J, Sagan C, Pere M, Chelha R, Olivier PY, Simon G, Rougon M, Pene F, Ferre A, Kamel T, Boyer A, Badie J, Hayon J, Decavele M, Garcon P, Richard JC, Argaud L, Hraiech S, Auchabie J, Foucault C, Legay F, Chanareille PM, Souweine B, Geri G, Delbove A, Bonny V, Beuret P, Vimpere D, Plantefeve G, Canet E. Post-mortem lung biopsies in fatal Covid-19 acute respiratory distress syndrome: a prospective cohort study of 169 patients (HISTOCOVID). Ann Intensive Care. 2025 Jun 11;15(1):80. doi: 10.1186/s13613-025-01493-5. PMID 40498264